CLINICAL TRIAL: NCT02895373
Title: A Prospective Randomized, Double Blind Study on Safety and Efficacy of Alprostadil as Additional Anticoagulant in Patients With Veno- Venous Extracorporeal Membrane Oxygenation (ECMO)
Brief Title: PGE1 as Additive Anticoagulant in ECMO-Therapy
Acronym: ECMO_PGE1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After completion of pilot study (n=50) no effect on primary outcome and limited feasibility of recruitment and study procedures
Sponsor: Thomas Staudinger (Other)
Responsible Party: Sponsor-Investigator, Thomas Staudinger, Ao.Univ.Prof. Dr. med, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ECMO_PGE1_2.1
Record Dates: First submitted 2016-06-30; First posted 2016-09-09 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-01

CONDITIONS: Respiratory Distress Syndrome, Adult; Extracorporeal Membrane Oxygenation
Keywords: platelet inhibition; alprostadil; extracorporeal membrane oxygenation; bleeding; thromboembolic
MeSH Terms: conditions — Respiratory Distress Syndrome; Hemorrhage | interventions — Alprostadil; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alprostadil (Experimental): heparin (dose adjusted to aptt 50-60s) + Alprostadil (=PGE1) 5ng/kg/min, continuously, start within 24h of initiation of ECMO therapy and end at the end of ECMO therapy
  Interventions: Drug: Alprostadil
- Placebo (Placebo Comparator): heparin (dose adjusted to aptt 50-60s) + 0.9% sodium chloride infusion, continuously, start within 24h of initiation of ECMO therapy and end at the end of ECMO therapy
  Interventions: Drug: 0.9% sodium chloride solution

INTERVENTIONS:
Drug: Alprostadil — 5ng/kg/min, continuously, start within 24h of initiation of ECMO therapy and end at the end of ECMO therapy
  Arms: Alprostadil
Drug: 0.9% sodium chloride solution — continuously, start within 24h of initiation of ECMO therapy and end at the end of ECMO therapy
  Arms: Placebo

SUMMARY:
Bleeding complications and thromboembolic complications are frequent during extracorporeal membrane oxygenation (ECMO). Retrospective data suggest that platelet inhibition using prostaglandins, in this case PGE1, may reduce thromboembolic complications without increasing the bleeding risk. This randomized, double-blind trial aims to investigate the effects of PGE1 on bleeding risk, thromboembolic complications and the function of the ECMO.

DETAILED DESCRIPTION:
Prostaglandins may inhibit platelet activation via the P2Y1 ADP receptor. Platelets may contribute to thromboembolic complications and coagulation activation during ECMO therapy. Retrospective data suggest that treatment with PGE1 may serve beneficial by reducing the amount of heparin needed for inhibition of coagulation activation, and by reducing the thromboembolic risk without increasing the risk of bleeding.

Inhibition of platelets via PGE1 (Alprostadil) may be interesting in this setting, because, in contrast to other platelet inhibitors, it has a very short half-life and platelets remain susceptible for activation by more potent agonists (i.e. thrombin, ADP). Thus, although reducing the contribution of platelets to coagulation activation, it may not affect safety of participating subjects.

This randomized, double-blind, placebo controlled trial will investigate whether treatment of patients with ECMO therapy proves beneficial.

ELIGIBILITY:
Inclusion Criteria:

* minimum age 18 years

  * Veno-Venous- ECMO
  * Minimum of 24h planned ECMO- therapy

Exclusion Criteria:

* • Long- term therapy with other antiplatelet drugs including Acetyl Salicylic Acid

  * known Heparin induced thrombocytopenia
  * Bleeding diathesis = contraindication for heparin (e.g. GI-bleeding, Intracerebral bleeding)
  * Platelets < 50 G/L
  * Thromboplastin time < 50%
  * Pregnancy
  * Patient < 18 years
  * prothrombin time <50%

Drop out criteria:

* Major bleeding (from Type 3 bleeding; see "primary objective")
* Occurrence of HIT (4 T- Score: Number of platelets, development over time, manifestation of thrombosis, other reasons for thrombocytopenia [10])
* Plt < 50 G/l

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Bleeding rate (quantified by the number of packed red blood cells transfused in relation to the duration of ECMO therapy) | up to 6 months
  The bleeding rate will be quantified by the number of packed red blood cells in relation to the duration of ECMO therapy. This duration may vary and cannot be predicted. Thus, we will calculate the required number of packed red blood cells i.e. per week.

SECONDARY OUTCOMES:
number of bleeding incidences and severity of bleeding (bleeding grades) | up to six months
  type 0: no bleeding type1: bleeding that is not actionable type 2: any overt actionable sign of hemorrhage type3: a) overt bleeding plut hb drop of 3-5g/dl b) >5g/dl, cardiac tamponade, requiring surgical intervention, bleeding requiring vasoactive agents c)intracranial bleeding, type 5: fatal bleeding
  number and severity of bleeding relative to the duration of ECMO therapy
Number of Clotting Events | up to six months
  * clinically noticeable thromboembolic events
  * cannulized veins (Duplex 24h after canula removal)
  * need of Membrane- changes,, macroscopic thrombus, discoloration
  * Global clotting tests (prothrombin time, activated partial thromboplastin time, Fibrinogen, D-Dimer)
  number of Clotting events in relation to the duration of ECMO therapy.
Function of the membrane oxygenator | up to six months
  The function of the membrane oxygenator will be assessed on a daily basis as part of clinical routine.This includes the capacity of oxygen transfer and carbon-dioxide (CO2) transfer.
Number of changes of the membrane oxygenator relative to the duration of ECMO therapy | up to six months
  Membrane oxygenators need to be changed due to loss of function (cause by clotting etc.).
Inflammation specific biomarkers (i.e. C-reactive protein, blood counts, reticulated platelets, etc.) | Time points: Immediately prior to initiation of ECMO, 24, 48 and 72h after initiation of ECMO, then twice a week until end of ECMO therapy, up to 12 months
  daily routine measurements and frozen plasma
Global Coagulation assays | Time points: Immediately prior to initiation of ECMO, 24, 48 and 72h after initiation of ECMO, then twice a week until end of ECMO therapy, up to 12 months
Thromboelastometry | Time points: Immediately prior to initiation of ECMO, 24, 48 and 72h after initiation of ECMO, then twice a week until end of ECMO therapy, up to 12 months
platelet function analyzer-100 | Time points: Immediately prior to initiation of ECMO, 24, 48 and 72h after initiation of ECMO, then twice a week until end of ECMO therapy, up to 12 months
Fibrinogen levels | Time points: Immediately prior to initiation of ECMO, 24, 48 and 72h after initiation of ECMO, then twice a week until end of ECMO therapy, up to 12 months
whole blood aggregometry | Time points: Immediately prior to initiation of ECMO, 24, 48 and 72h after initiation of ECMO, then twice a week until end of ECMO therapy, up to 12 months
D-Dimer levels | Time points: Immediately prior to initiation of ECMO, 24, 48 and 72h after initiation of ECMO, then twice a week until end of ECMO therapy, up to 12 months
Catecholamines | Time points: Immediately prior to initiation of ECMO, 24, 48 and 72h after initiation of ECMO, then twice a week until end of ECMO therapy, up to 12 months
  need for and dose of catecholamines
cardiac output | Time points: Immediately prior to initiation of ECMO, 24, 48 and 72h after initiation of ECMO, then twice a week until end of ECMO therapy, up to 12 months
blood pressure | Time points: Immediately prior to initiation of ECMO, 24, 48 and 72h after initiation of ECMO, then twice a week until end of ECMO therapy, up to 12 months
mortality | Day 28/90, ICU mortality assessed at the discharge from the Intensive Care unit, this will be up to 12 months after inclusion into the study
  by chart review or telephone call
number of platelet transfusions, fresh frozen plamsa, coagulation interventions etc. | up to six months
  by chart review, number relative to the duration of ECMO therapy
number of platelet transfusions | up to six months
  by chart review, number relative to the duration of ECMO therapy
number of coagulation interventions | up to six months
  by chart review, number relative to the duration of ECMO therapy

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Staudinger, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Department of Medicine I, Intensive Care Unit, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No
Data will be published in a peer-reviewed journal, individual data will not be made publicly available except by a direct request to the PI (in an anonymized fashion)

REFERENCES:
- [Derived] Buchtele N, Schorgenhofer C, Schwameis M, Jilma B, Schellongowski P, Herkner H, Riss K, Schmid M, Hermann A, Robak O, Nagler B, Traby L, Bojic A, Staudinger T. Add-On Prostaglandin E1 in Venovenous Extracorporeal Membrane Oxygenation: A Randomized, Double-Blind, Placebo-controlled Pilot Trial. Am J Respir Crit Care Med. 2022 Jul 15;206(2):170-177. doi: 10.1164/rccm.202110-2359OC. PMID 35426776